CLINICAL TRIAL: NCT06923631
Title: Unravelling the Measles Paradox in Children: a Disease Associated With Both Immune Suppression and Immune Activation
Brief Title: Unravelling the Measles Paradox in Children
Acronym: MISIA-k
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Corine Geurts van Kessel, Medical microbiologist, Erasmus Medical Center
Other Study IDs: NL-009458
Record Dates: First submitted 2025-03-27; First posted 2025-04-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: MEASLES DISEASE
Keywords: measles; immune response
MeSH Terms: conditions — Measles

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10mL of whole blood, 1 throat swab and 1 nasal fluid lining collector (nasosorption) per study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (max 50 inclusions): Unprotected children with at least one sibling diagnosed with measles
- Group B (max 50 inclusions): Age matched children with detectable immunity to MeV

SUMMARY:
Measles is caused by measles virus (MeV). The disease is associated with lymphopenia and immune suppression, which is an important cause of measles-associated morbidity and mortality. Measles-induced immune suppression can last several years, whereas measles lymphopenia is usually resolved within two weeks. At the same time, measles induces lifelong immunity. This apparent contradiction, known as the 'measles paradox', was partially solved when investigators demonstrated that MeV infects and depletes pre-existing memory cells, thereby causing 'immune amnesia'. This model is supported by observations in animal models and clinical studies, but several questions remain to be addressed, like the duration of measles-induced amnesia and changes in the immune repertoire after measles. to address the immunological questions regarding MeV infection.

DETAILED DESCRIPTION:
Measles is caused by measles virus (MeV). The disease is associated with lymphopenia and immune suppression, which is an important cause of measles-associated morbidity and mortality. Measles-induced immune suppression can last several years, whereas measles lymphopenia is usually resolved within two weeks. At the same time, measles induces lifelong immunity. This apparent contradiction, known as the 'measles paradox', was partially solved when investigators demonstrated that MeV infects and depletes pre-existing memory cells, thereby causing 'immune amnesia'. This model is supported by observations in animal models and clinical studies, but several questions remain to be addressed, like the duration of measles-induced amnesia and changes in the immune repertoire after measles. Recently, investigators have acquired permission to address these remaining questions in 18-25 years old adults (MEC-2024-0230). However, investigators have reservations about the feasibility of including enough participants between 18 and 25 years old that have not been vaccinated against or infected with MeV; it is possible that investigators will not reach sufficient inclusions to address the immunological questions regarding MeV infection in that protocol. Therefore, investigators propose to additionally study these questions in children in the age of 4 up to and including 17.

ELIGIBILITY:
Inclusion Criteria:

Group A

* Aged 4 - 17 years old
* Susceptible to measles
* No pre-existing immunity against measles (vaccination or earlier infection)

Group B

* Aged 4 - 17 years old
* Protected against measles due to vaccination or earlier infection

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Diagnosed chronic disease that lasted over 3 months
* Immune suppression (due to medication or underlying disease)
* Group A; Detectable MeV-antibodies in the T1 blood sample

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in group A will be from 4 up to and including 17 years of age and include children who are not protected against measles. Families willing to participate will self-identify them to the researchers, with the help of schools, Municipal Health Services and regional general practitioners.
  Children in group B will be from 4 up to and including 17 years of age and have received one or two MMR vaccinations, depending on their age. The children will be recruited from the same geographical regions with low vaccine coverage as the children in group A, for example classmates.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Compare measles-induced loss of pathogen-specific antibodies | 36 months
  The investigators will measure changes in the immune repertoire using longitudinal samples obtained from children who are infected with MeV. To this end, they will measure pathogen-specific antibody responses (titers) pre- and post-measles and compare these to determine whether measles led to a loss of pathogen-specific antibodies.
Compare measles-induced loss of pathogen-specific T-cells | 36 months
  The investigators will measure changes in the immune repertoire using longitudinal samples obtained from children who are infected with MeV. To this end, they will measure pathogen-specific T-cell responses (frequencies) pre- and post-measles and compare these to determine whether measles led to a loss of pathogen-specific T-cells.

CONTACTS AND LOCATIONS:
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Velzen E, de Coster E, van Binnendijk R, Hahne S. Measles outbreak in an anthroposophic community in The Hague, The Netherlands, June-July 2008. Euro Surveill. 2008 Jul 31;13(31):18945. No abstract available. PMID 18761905
- [Background] Mollema L, Harmsen IA, Broekhuizen E, Clijnk R, De Melker H, Paulussen T, Kok G, Ruiter R, Das E. Disease detection or public opinion reflection? Content analysis of tweets, other social media, and online newspapers during the measles outbreak in The Netherlands in 2013. J Med Internet Res. 2015 May 26;17(5):e128. doi: 10.2196/jmir.3863. PMID 26013683
- [Background] Laksono BM, de Vries RD, Verburgh RJ, Visser EG, de Jong A, Fraaij PLA, Ruijs WLM, Nieuwenhuijse DF, van den Ham HJ, Koopmans MPG, van Zelm MC, Osterhaus ADME, de Swart RL. Studies into the mechanism of measles-associated immune suppression during a measles outbreak in the Netherlands. Nat Commun. 2018 Nov 23;9(1):4944. doi: 10.1038/s41467-018-07515-0. PMID 30470742
- [Background] Knol M, Urbanus A, Swart E, Mollema L, Ruijs W, van Binnendijk R, Te Wierik M, de Melker H, Timen A, Hahne S. Large ongoing measles outbreak in a religious community in the Netherlands since May 2013. Euro Surveill. 2013 Sep 5;18(36):pii=20580. doi: 10.2807/1560-7917.es2013.18.36.20580. PMID 24079377
- [Background] Van Den Hof S, Smit C, Van Steenbergen JE, De Melker HE. Hospitalizations during a measles epidemic in the Netherlands, 1999 to 2000. Pediatr Infect Dis J. 2002 Dec;21(12):1146-50. doi: 10.1097/00006454-200212000-00012. PMID 12488666
- [Background] Mina MJ, Kula T, Leng Y, Li M, de Vries RD, Knip M, Siljander H, Rewers M, Choy DF, Wilson MS, Larman HB, Nelson AN, Griffin DE, de Swart RL, Elledge SJ. Measles virus infection diminishes preexisting antibodies that offer protection from other pathogens. Science. 2019 Nov 1;366(6465):599-606. doi: 10.1126/science.aay6485. PMID 31672891
- [Background] Rennick LJ, de Vries RD, Carsillo TJ, Lemon K, van Amerongen G, Ludlow M, Nguyen DT, Yuksel S, Verburgh RJ, Haddock P, McQuaid S, Duprex WP, de Swart RL. Live-attenuated measles virus vaccine targets dendritic cells and macrophages in muscle of nonhuman primates. J Virol. 2015 Feb;89(4):2192-200. doi: 10.1128/JVI.02924-14. Epub 2014 Dec 3. PMID 25473055
- [Background] de Vries RD, Lemon K, Ludlow M, McQuaid S, Yuksel S, van Amerongen G, Rennick LJ, Rima BK, Osterhaus AD, de Swart RL, Duprex WP. In vivo tropism of attenuated and pathogenic measles virus expressing green fluorescent protein in macaques. J Virol. 2010 May;84(9):4714-24. doi: 10.1128/JVI.02633-09. Epub 2010 Feb 24. PMID 20181691
- [Background] Aaby P, Bukh J, Lisse IM, Smits AJ. Measles vaccination and reduction in child mortality: a community study from Guinea-Bissau. J Infect. 1984 Jan;8(1):13-21. doi: 10.1016/s0163-4453(84)93192-x. PMID 6699411
- [Background] Sato R, Haraguchi M. Effect of measles prevalence and vaccination coverage on other disease burden: evidence of measles immune amnesia in 46 African countries. Hum Vaccin Immunother. 2021 Dec 2;17(12):5361-5366. doi: 10.1080/21645515.2021.2013078. Epub 2021 Dec 29. PMID 34965183
- [Background] Petrova VN, Sawatsky B, Han AX, Laksono BM, Walz L, Parker E, Pieper K, Anderson CA, de Vries RD, Lanzavecchia A, Kellam P, von Messling V, de Swart RL, Russell CA. Incomplete genetic reconstitution of B cell pools contributes to prolonged immunosuppression after measles. Sci Immunol. 2019 Nov 1;4(41):eaay6125. doi: 10.1126/sciimmunol.aay6125. PMID 31672862
- [Background] Cox RM, Wolf JD, Lieberman NA, Lieber CM, Kang HJ, Sticher ZM, Yoon JJ, Andrews MK, Govindarajan M, Krueger RE, Sobolik EB, Natchus MG, Gewirtz AT, deSwart RL, Kolykhalov AA, Hekmatyar K, Sakamoto K, Greninger AL, Plemper RK. Therapeutic mitigation of measles-like immune amnesia and exacerbated disease after prior respiratory virus infections in ferrets. Nat Commun. 2024 Feb 8;15(1):1189. doi: 10.1038/s41467-024-45418-5. PMID 38331906
- [Background] Laksono BM, Roelofs D, Comvalius AD, Schmitz KS, Rijsbergen LC, Geers D, Nambulli S, van Run P, Duprex WP, van den Brand JMA, de Vries RD, de Swart RL. Infection of ferrets with wild type-based recombinant canine distemper virus overwhelms the immune system and causes fatal systemic disease. mSphere. 2023 Aug 24;8(4):e0008223. doi: 10.1128/msphere.00082-23. Epub 2023 Jun 28. PMID 37377421
- [Background] Ward BJ, Johnson RT, Vaisberg A, Jauregui E, Griffin DE. Cytokine production in vitro and the lymphoproliferative defect of natural measles virus infection. Clin Immunol Immunopathol. 1991 Nov;61(2 Pt 1):236-48. doi: 10.1016/s0090-1229(05)80027-3. PMID 1914259
- [Background] Hirsch RL, Griffin DE, Johnson RT, Cooper SJ, Lindo de Soriano I, Roedenbeck S, Vaisberg A. Cellular immune responses during complicated and uncomplicated measles virus infections of man. Clin Immunol Immunopathol. 1984 Apr;31(1):1-12. doi: 10.1016/0090-1229(84)90184-3. PMID 6230187
- [Background] Tamashiro VG, Perez HH, Griffin DE. Prospective study of the magnitude and duration of changes in tuberculin reactivity during uncomplicated and complicated measles. Pediatr Infect Dis J. 1987 May;6(5):451-4. doi: 10.1097/00006454-198705000-00007. PMID 3601492
- [Background] de Vries RD, McQuaid S, van Amerongen G, Yuksel S, Verburgh RJ, Osterhaus AD, Duprex WP, de Swart RL. Measles immune suppression: lessons from the macaque model. PLoS Pathog. 2012;8(8):e1002885. doi: 10.1371/journal.ppat.1002885. Epub 2012 Aug 30. PMID 22952446
- [Background] de Swart RL, Ludlow M, de Witte L, Yanagi Y, van Amerongen G, McQuaid S, Yuksel S, Geijtenbeek TB, Duprex WP, Osterhaus AD. Predominant infection of CD150+ lymphocytes and dendritic cells during measles virus infection of macaques. PLoS Pathog. 2007 Nov;3(11):e178. doi: 10.1371/journal.ppat.0030178. PMID 18020706
- [Background] Mina MJ, Metcalf CJ, de Swart RL, Osterhaus AD, Grenfell BT. Long-term measles-induced immunomodulation increases overall childhood infectious disease mortality. Science. 2015 May 8;348(6235):694-9. doi: 10.1126/science.aaa3662. Epub 2015 May 7. PMID 25954009
- [Background] Ludlow M, Lemon K, de Vries RD, McQuaid S, Millar EL, van Amerongen G, Yuksel S, Verburgh RJ, Osterhaus AD, de Swart RL, Duprex WP. Measles virus infection of epithelial cells in the macaque upper respiratory tract is mediated by subepithelial immune cells. J Virol. 2013 Apr;87(7):4033-42. doi: 10.1128/JVI.03258-12. Epub 2013 Jan 30. PMID 23365435
- [Background] Ludlow M, de Vries RD, Lemon K, McQuaid S, Millar E, van Amerongen G, Yuksel S, Verburgh RJ, Osterhaus ADME, de Swart RL, Duprex WP. Infection of lymphoid tissues in the macaque upper respiratory tract contributes to the emergence of transmissible measles virus. J Gen Virol. 2013 Sep;94(Pt 9):1933-1944. doi: 10.1099/vir.0.054650-0. Epub 2013 Jun 19. PMID 23784446
- [Background] Lemon K, de Vries RD, Mesman AW, McQuaid S, van Amerongen G, Yuksel S, Ludlow M, Rennick LJ, Kuiken T, Rima BK, Geijtenbeek TB, Osterhaus AD, Duprex WP, de Swart RL. Early target cells of measles virus after aerosol infection of non-human primates. PLoS Pathog. 2011 Jan 27;7(1):e1001263. doi: 10.1371/journal.ppat.1001263. PMID 21304593
- [Background] Laksono BM, de Vries RD, McQuaid S, Duprex WP, de Swart RL. Measles Virus Host Invasion and Pathogenesis. Viruses. 2016 Jul 28;8(8):210. doi: 10.3390/v8080210. PMID 27483301
- [Background] Laksono BM, de Vries RD, Duprex WP, de Swart RL. Measles pathogenesis, immune suppression and animal models. Curr Opin Virol. 2020 Apr;41:31-37. doi: 10.1016/j.coviro.2020.03.002. Epub 2020 Apr 24. PMID 32339942
- [Background] de Vries RD, de Swart RL. Measles immune suppression: functional impairment or numbers game? PLoS Pathog. 2014 Dec 18;10(12):e1004482. doi: 10.1371/journal.ppat.1004482. eCollection 2014 Dec. No abstract available. PMID 25522010
- See also: WHO measles factsheet — https://www.who.int/news-room/fact-sheets/detail/measles
- See also: A 30-fold rise of measles cases in 2023 in the WHO European Region warrants urgent action — https://www.who.int/europe/news-room/14-12-2023-a-30-fold-rise-of-measles-cases-in-2023-in-the-who-european-region-warrants-urgent-action
- See also: Threat assessment brief: Measles on the rise in the EU/EEA - Considerations for public health response — https://www.ecdc.europa.eu/en/publications-data/threat-assessment-brief-measles-rise-eueea-considerations-public-health-response